CLINICAL TRIAL: NCT01857037
Title: Detection and Localization of Prostate Cancer Local Recurrences After Radiation Therapy Using Histoscanning™ and Multiparametric MRI
Brief Title: Post-radiation Prostate Cancer Local Recurrences: Detection With Histoscanning™ and MRI
Acronym: HISTO-RAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010.655
Record Dates: First submitted 2012-03-28; First posted 2013-05-20 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): Single arm
  Interventions: Other: Histoscanning™ and multiparametric MRI

INTERVENTIONS:
Other: Histoscanning™ and multiparametric MRI — Detection and localization of prostate cancer local recurrences after radiation therapy using Histoscanning™ and multiparametric MRI

SUMMARY:
Inclusion criteria:

* Patients with biochemical recurrence (Phoenix criteria: PSA nadir + 2 ng/ml) after radiation therapy for prostate cancer addressed for prostate biopsy OR
* Patients referred to our institution for biopsy-proven local recurrence after radiation therapy for prostate cancer but needing a re-assessment with biopsy (insufficient number of biopsy and/or imprecise location of positive biopsy and/or questionable diagnostic of recurrence)

Study Design:

* Included patients will undergo an endorectal US examination with a Histoscanning™ acquisition and a multiparametric (T2-weighted, diffusion-weighted and dynamic contrast-enhanced) MRI.
* Two independent operators will separately define suspicious focal lesion on Histoscanning™ images and on MR images.
* Random biopsies (at least 2 cores) will be performed in sextants negative at Histoscanning™ and at MRI ; In sextants positive at Histoscanning™ and/or at MRI, targeted biopsies will be performed in the suspicious part of the sextant (at least two cores per suspicious lesion).
* Histoscanning™ and MRI results will be compared to biopsy results.

A total of 30 patients will be included

ELIGIBILITY:
Inclusion Criteria:

* Patients with biochemical recurrence (Phoenix criteria: PSA nadir + 2 ng/ml) after radiation therapy for prostate cancer addressed for prostate biopsy OR Patients referred to our institution for biopsy-proven local recurrence after radiation therapy for prostate cancer but needing a re-assessment with biopsy (insufficient number of biopsy and/or imprecise location of positive biopsy and/or questionable diagnostic of recurrence)
* IRB-approved informed consent signed

Exclusion Criteria:

* Contraindication to MRI
* Contraindication to endorectal examination
* Contraindication to prostate biopsy
* History of allergy to gadolinium chelates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of Histoscanning™ after radiation therapy in comparison to random and targeted biopsy. | 1 day
  Histoscanning and biopsy findings will be compared on a sextant by sextant basis. A mixed effects logistic regression model (with fixed and random effects) will be used to model the sensitivity and specificity of Histoscanning to correctly identify the presence or absence of cancer into prostate sextants.

SECONDARY OUTCOMES:
Evaluation of multiparametric MRI after radiation therapy in comparison to random and targeted biopsy. | 1 day
  MRI and biopsy findings will be compared on a sextant by sextant basis. A mixed effects logistic regression model (with fixed and random effects) will be used to model the sensitivity and specificity of MRI to correctly identify the presence or absence of cancer into prostate sextants.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rouvière, Pr, Principal Investigator — Hospices Civiles de Lyon
Locations (1):
- Prof O. ROUVIERE, Lyon, Rhône, France

REFERENCES:
- [Background] Alonzo F, Melodelima C, Bratan F, Vitry T, Crouzet S, Gelet A, Rouviere O. Detection of locally radio-recurrent prostate cancer at multiparametric MRI: Can dynamic contrast-enhanced imaging be omitted? Diagn Interv Imaging. 2016 Apr;97(4):433-41. doi: 10.1016/j.diii.2016.01.008. Epub 2016 Feb 23. PMID 26928245